CLINICAL TRIAL: NCT02744885
Title: Crave Crush: Sugar Cravings and ad Lib Candy Uptake
Brief Title: Crave Crush Behavioral Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oregon Research Behavioral Intervention Strategies, Inc. (Industry)
Collaborators: Cravecrush (Unknown); Oregon Behavioral Intervention Strategies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: FOUR001
Record Dates: First submitted 2016-04-18; First posted 2016-04-20 (Estimated); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Crave Crush (Experimental): Crave Crush is a plant-based tablet that alters taste perception by affecting sweet taste receptors on the tongue.
  Interventions: Dietary Supplement: Crave Crush
- Placebo (Placebo Comparator): The placebo tablet is comparable in taste and is comprised primarily of sorbitol.
  Interventions: Dietary Supplement: Placebo Comparator: Placebo

INTERVENTIONS:
Dietary Supplement: Crave Crush — Crave Crush is a dietary supplement that affects sweet taste receptors on the tongue.
  Arms: Crave Crush
Dietary Supplement: Placebo Comparator: Placebo — The placebo tablet is comparable in taste and is comprised primarily of sorbitol.
  Arms: Placebo

SUMMARY:
The purpose of the research is to determine if participants who take "Crave Crush" will report lower cravings and palatability ratings of candy as compared to subjects who receive the placebo. Participants are self-selected university students who pass our table and verbally agree to participate in a research study about taste preferences. Data will be recorded anonymously.

DETAILED DESCRIPTION:
When students approach the table, research assistants will ask them to choose their favorite kind of candy from an assortment. They will ask the subjects to rate their craving for the candy before they taste it. After they try the candy, the research assistants will ask them to rate its palatability. Then they will rate their craving for another piece of candy. A research assistant will flip a coin to determine whether the subject will receive Crave Crush or placebo. While the Crave Crush or placebo is dissolving in the mouth, the students will fill out a short questionnaire with an identification number. The questionnaire will ask for their age, gender, ethnicity, approximate height and weight, and a few questions about their dietary habits.

After the tablet dissolves, research assistants will ask the students to rate their craving for another piece of candy. Research assistants will ask participants if they would like another piece of candy and have them assess palatability again. The process of offering a piece of candy and asking subjects to rate palatability will occur up to five times. Finally, subjects will be asked if they would like to take a few pieces of candy for the road and if they say yes, the number of pieces they take with them will be noted. The study activities should last no more than 5-10 minutes per participant.

ELIGIBILITY:
Inclusion Criteria:

* University student, having eaten within the last hour, having slept within two hours of their normal amount

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2016-02; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Self-Reported Craving Reduction | 10 minutes

SECONDARY OUTCOMES:
Self-Reported Palatability Reduction | 10 minutes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stice E, Yokum S, Gau JM. Gymnemic acids lozenge reduces short-term consumption of high-sugar food: A placebo controlled experiment. J Psychopharmacol. 2017 Nov;31(11):1496-1502. doi: 10.1177/0269881117728541. Epub 2017 Sep 25. PMID 28944714